CLINICAL TRIAL: NCT07238660
Title: A Randomized Controlled Trial Comparing Thoracic Expansion Exercises and Dynamic Neuromuscular Stabilization on Respiratory Function and Bilateral Trapezius Muscle Activity in Individuals With Forward Head Posture
Brief Title: Thoracic Expansion vs DNS Exercises in Forward Head Posture
Acronym: FHP-DNS-TE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra BECENI (Other)
Responsible Party: Sponsor-Investigator, Esra BECENI, lecturer, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-FHP-DNS-TE-2025-01
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Forward Head Posture
Keywords: craniovertebral angle; respiratory function test; electromyography; Dynamic Neuromuscular Stabilization(DNS); breathing exercises

STUDY DESIGN:
Intervention Model Description: a randomized, controlled, assessor-blind, prospective study
Who Masked: Outcomes Assessor
Masking Description: Randomization will be done by the sealed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Neuromuscular Stabilization Group (DNSG) (Experimental): Developmental DNS patterns (supine 90/90, prone on elbows, quadruped), performed twice daily for 6 weeks.
  Interventions: Behavioral: Dynamic Neuromuscular Stabilization Exercises
- Thoracic Expansion Exercise Group (TEG) (Experimental): Upper, middle, and lower lobe-focused thoracic expansion breathing exercises, twice daily for 6 weeks.
  Interventions: Behavioral: Thoracic Expansion Exercise

INTERVENTIONS:
Behavioral: Dynamic Neuromuscular Stabilization Exercises — Participants in the DNS group will perform Dynamic Neuromuscular Stabilization exercises based on developmental kinesiology principles. The program consists of three standardized DNS patterns:
  Supine 90°/90° Position (4.5-month developmental stage): The participant lies supine with hips and knees flexed to 90°, emphasizing diaphragmatic breathing, rib cage expansion, and neutral spine alignment.
  Prone on Elbows (4.5-month stage): The participant supports the upper body on elbows while maintaining cervical neutrality and coordinated diaphragmatic breathing.
  Quadruped Position (9-month developmental stage): The participant maintains a four-point kneeling position with proper spinal stabilization and controlled breathing.
  All exercises focus on coordinated activation of deep cervical flexors, diaphragm, transversus abdominis, multifidus, and pelvic floor muscles.
  Participants will perform 2 supervised sessions per week and twice-daily home exercises (10 repetitions × 3 sets) for 6 weeks.
  Arms: Dynamic Neuromuscular Stabilization Group (DNSG)
Behavioral: Thoracic Expansion Exercise — Participants in the thoracic expansion group will perform a structured breathing exercise program focused on increasing upper, middle, and lower thoracic mobility. The program includes:
  Upper Lobe Expansion Exercise: Participant places hands over upper thoracic region and performs deep inhalation to expand upper lung fields, followed by slow exhalation.
  Middle Lobe Expansion Exercise: Hands placed laterally at mid-thoracic level to facilitate expansion of the middle lobes during inhalation.
  Lower Lobe Expansion Exercise: Hands positioned over the lower rib cage to promote diaphragmatic and lower thoracic expansion.
  Each exercise is performed for 3 sets of 10 repetitions, twice daily, for 6 weeks. Two supervised sessions per week will ensure correct technique and progression. The exercises aim to improve thoracic mobility, respiratory mechanics, and chest wall expansion.
  Arms: Thoracic Expansion Exercise Group (TEG)

SUMMARY:
This randomized controlled trial aims to compare the effects of thoracic expansion exercises and Dynamic Neuromuscular Stabilization (DNS) on respiratory function and bilateral trapezius muscle activity in individuals with forward head posture (FHP). A total of 32 participants aged 18-40 years with a craniovertebral angle (CVA) of less than 53° will be randomly assigned to either the DNS group or the thoracic expansion exercise group. Primary outcomes include respiratory function (FEV1, FVC, FEV1/FVC), trapezius muscle activation measured with EMG biofeedback, and craniovertebral angle. Secondary outcomes include thoracic mobility and health-related quality of life assessed using the St. George's Respiratory Questionnaire. Both interventions will be applied for 6 weeks. The study aims to determine which approach provides greater improvement in posture-related respiratory dysfunction and muscle activation.

DETAILED DESCRIPTION:
Forward head posture (FHP) is a common postural deviation characterized by reduced craniovertebral angle (CVA), altered cervicothoracic alignment, and compensatory activation of accessory respiratory muscles. Individuals with FHP frequently demonstrate limited thoracic mobility, decreased respiratory efficiency, and increased demand on superficial neck musculature. These biomechanical alterations may negatively influence pulmonary function parameters such as FEV1 and FVC, as well as contribute to elevated electromyographic (EMG) activity in the upper trapezius muscles.

Various therapeutic approaches have been developed to address posture-related respiratory dysfunction. Thoracic expansion breathing exercises aim to enhance chest wall mobility and improve lung expansion across upper, middle, and lower thoracic regions. Dynamic Neuromuscular Stabilization (DNS), based on developmental kinesiology principles, seeks to optimize diaphragmatic function, intra-abdominal pressure regulation, and coordinated activation of deep stabilizing musculature. Although both methods have theoretical benefits for improving respiratory mechanics and postural alignment, comparative evidence regarding their differential effects in individuals with FHP remains limited.

This randomized controlled trial will investigate the immediate and short-term effects of thoracic expansion breathing exercises versus DNS-based stabilization exercises on respiratory function, cervicothoracic posture, and muscle activation patterns. Thirty-two adults aged 18-40 years with a CVA of less than 53° will be enrolled and randomly assigned using an opaque envelope method to one of two intervention groups: the Thoracic Expansion Exercise Group or the Dynamic Neuromuscular Stabilization Group. Each intervention protocol will be implemented over a 6-week period, consisting of twice-weekly supervised sessions complemented by twice-daily home exercise routines.

Outcome assessments will be conducted at baseline and at the end of the 6-week intervention period. These assessments will include: CVA measured by standardized lateral photography and ImageJ analysis; bilateral upper trapezius muscle activity assessed using surface EMG biofeedback; pulmonary function tests (FEV1, FVC, FEV1/FVC) conducted with spirometry; thoracic expansion measured at three levels using a tape-measure chest mobility test; and health-related quality of life evaluated with the St. George's Respiratory Questionnaire (SGRQ). The study protocol was approved by the Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee.

This trial is designed to provide a comparative analysis of two commonly used physiotherapy interventions for FHP, with a focus on their effects on posture-related respiratory mechanics, thoracic mobility, and neuromuscular activation. All findings will be reported separately in the Results section. The present description outlines the scientific rationale, study design, and intervention procedures without duplicating eligibility criteria or outcome measure definitions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 40 years.
* Craniovertebral angle (CVA < 53°) indicating forward head posture.
* Able to perform exercise-based interventions.
* Voluntarily agrees to participate and signs the informed consent form.
* No neurological, orthopedic, systemic, or cardiopulmonary conditions that would limit participation.

Exclusion Criteria:

* Contraindications to exercise (e.g., acute musculoskeletal injury, uncontrolled cardiovascular disease).
* Chronic upper respiratory tract disease that may affect spirometry results. Presence of a cardiac pacemaker.
* Neurological disorders, systemic diseases, or mental impairments that could interfere with exercise cooperation.
* History of orthopedic or musculoskeletal surgery affecting mobility or posture.
* Currently participating in respiratory exercises, spinal stabilization training, or structured exercise programs.
* Engagement in professional sports or intensive physical training that may affect baseline neuromuscular measurements.
* Failure to comply with the exercise program (e.g., missing 3 consecutive days of prescribed exercises).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) | Baseline and Week 6
  CVA is used to assess forward head posture. Participants will be asked to stand in a natural and relaxed posture while focusing on a marked point at eye level on the wall. A lateral photograph will be taken using a Iphone 13 camera mounted on a tripod at shoulder height and placed 1.5 meters from the participant. The spinous process of the C7 vertebra and the tragus of the ear will be marked. The angle between the line connecting the tragus to C7 and a horizontal reference line will be calculated using the ImageJ software. The measurement results will be recorded on the evaluation form.
  Analysis Metric: Change in CVA (degrees)

SECONDARY OUTCOMES:
Trapezius Muscle Activity (Surface EMG Biofeedback, µV) | Baseline and Week 6
  Surface EMG sensors will be placed bilaterally over the upper trapezius muscles. Participants will perform three 5-second isometric contractions, and the mean amplitude (µV) of the signals will be recorded.
  Analysis metric: Change from baseline to Week 6 in mean EMG amplitude of bilateral upper trapezius
FEV1 (Forced Expiratory Volume in 1 Second) | Baseline and Week 6
  FEV1 will be recorded using a portable spirometer (BTL-08 Spiro Pro). The highest value of three acceptable forced expiratory maneuvers will be used.
  Analysis Metric: Change from baseline to Week 6 (liters)
FVC (Forced Vital Capacity) | Baseline and Week 6
  FVC will be assessed using standard spirometry procedures. Three maximal forced expiratory maneuvers will be performed, and the best value will be recorded.
  Analysis Metric:
  Change from baseline to Week 6 (liters)
Thoracic Expansion (Chest Mobility, cm) | Baseline and Week 6
  Thoracic expansion will be measured with a tape measure at upper, middle, and lower thoracic levels. The difference between maximum inhalation and exhalation will be used as the thoracic mobility value.
  Analysis Metric:
  Change from baseline to Week 6 (cm)
St. George's Respiratory Questionnaire (SGRQ) Total Score | Baseline and Week 6
  The SGRQ is a standardized instrument assessing symptoms, activity limitation, and psychosocial impact related to respiratory dysfunction. Scores range from 0 to 100, with higher scores indicating worse health status and greater impairment.
  Analysis Metric:
  Change from baseline to Week 6 (0-100 score)

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Yalçın, PhD, Study Director — Mudanya University, Faculty of Health Sciences, Department of Physiotherapy; Esra Beceni, Lecturer, Principal Investigator — Mudanya University Vocational, Physiotherapy Program
Locations (1):
- Mudanya University, Bursa, Turkey (Türkiye)